CLINICAL TRIAL: NCT03357354
Title: Program for Screening and Prevention of Eating Disorders in Obese Young People in Vulnerable Neighborhoods of Marseille: an Action Research
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty of inclusion
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-31
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2017-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obese Children in precarious situations (Experimental)
  Interventions: Behavioral: collective workshop

INTERVENTIONS:
Behavioral: collective workshop — diet, sports games, food budget, feeling of satiety and hunger, self-image

SUMMARY:
Action research has been developed in this direction in order to use a tool to identify food disorder behavior among obese youths in their neighborhoods and social centers in vulnerable neighborhoods of Marseille, with the aim of a multi-professional therapeutic management (psychosocial support, theater) and a specialized orientation.

This program consists of the participation of each patient recruited in collective workshops. A total of 60 patients considered. Our hypothesis lies in the fact that for young people to participate in an adapted device, taking into account the global needs of young people and their entourage, would limit the deleterious effects of obesity and promote the young person's autonomy and allow him to be a actor in the request for care.

The project's objective is to provide support in the form of workshops with patients identified by the Marseille Hospitals Public Assistance Health Center as obese children and adolescents, in a precarious situation; to identify the presence of binge eating disorders and evaluate the impact of participation in these workshops on subsequent management by highly specialized professionals in food disorder behavior.

DETAILED DESCRIPTION:
The mobile team (EM) of the Marseille Hospitals Public Assistance Health Center has the mission to inform, screen, support and guide the access to care of people in targeted neighborhoods, said to be vulnerable, by the city's policy of Marseille. The health space, a place of welcome and care, is located at a distance from any hospital structure within the most vulnerable neighborhoods of the city.

ELIGIBILITY:
Inclusion Criteria :

* Boys or girls aged 11 to 17
* Reside in the territory of intervention of the mobile team, i.e the 3rd, 14th, 15th and 16th arrondissement of Marseille, districts said to be vulnerable by the city's policy.
* Body mass index greater than or equal to IOTF-30 (HAS, 2011)
* Social precariousness score EPICES greater than or equal to 30riteria:
* Diagnosed Eating Disorder without medical and/or multi-professional care

Exclusion Criteria:

* Child with major difficulty of behavior
* Patient with medical care

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Number of subjects included in the three months following the end of the workshops in a device specialized in the management of behavioral disorders. | 6 MONTHS
  Tracking interview after the end of workshops

SECONDARY OUTCOMES:
Evaluation of with the ADO-BEDS | 6 MONTHS
  children and teenagers will be asked to answer some items

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France